CLINICAL TRIAL: NCT02083211
Title: Phase III Clinical Trial: "Evaluation of the Combination of Nimotuzumab and Cisplatin-Vinorelbine in First Line Chemotherapy in the Survival of Patients With Recurring-Persistent Cervical Carcinoma"
Brief Title: Combination of Nimotuzumab Cisplatin-Vinorelbine in First Line Chemotherapy in Recurring-Persistent Cervical Carcinoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Cancerología (Other Government)
Collaborators: Laboratorios Pisa S.A. de C.V. (Industry); National Heart Institute, Mexico (Other Government)
Responsible Party: Principal Investigator, Dr. Lucely Cetina Pérez, MsC, MD, National Institute of Cancerología
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NIMO 001-09 MX
Record Dates: First submitted 2014-02-17; First posted 2014-03-11 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Cervical Cancer Recurrent or Persistent; Palliative Treatment; Monoclonal Antibody in Cervical Cancer Treatment
Keywords: Cervical cancer; Recurrent or persistent tumor; Monoclonal antibody
MeSH Terms: conditions — Uterine Cervical Neoplasms; Recurrence

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- mAb Nimotuzumab + chemotherapy (Experimental)
  Interventions: Drug: mAb Nimotuzumab
- placebo + chemotherapy (Placebo Comparator)
  Interventions: Device: Placebo

INTERVENTIONS:
Drug: mAb Nimotuzumab — This group will receive a dose of 200 mg mAb hR3 (weekly over 18 weeks) plus chemotherapy (6 cycles every 21 days of Cisplatin (CDDP) 50 mg/m2 on day 1/, Vinorelbine 30 mg/m2 on day 1 and day 8)
  Arms: mAb Nimotuzumab + chemotherapy
Device: Placebo — This group will receive a placebo in addition to chemotherapy in a similar regimen. Once the chemotherapy is completed a maintenance dose will be administered with 200 mg/dose of mAb hR3 every 14 days until progression.
  Arms: placebo + chemotherapy

SUMMARY:
This study evauates the global survival of patients following administration of mAb Nimotuzumab hR3 + chemotherapy in the treatment of cervical cancer in first line therapy, after relapsing from chemo-radiotherapy.

It is a Phase III, multi-centric, randomized, double blind study; 168 patients will be assigned to Nimotuzumab + Cisplatin/Vinorelbine or placebo + Cisplatin/Vinorelbine. After progression, a second line chemotherapy based on carboplatino/taxol will be administered in both groups. Concomitant administration of Nimotuzumab will be continued every 14 days until limiting toxicity or ECOCG >3.

Tumor markers such as Kras, p53, KI67, and EGFR will be identified. Cardiac toxicity will be evaluated using MRI.

DETAILED DESCRIPTION:
Specific Objectives

1. To determine the global survival of patients treated with mAb Nimotuzumab hR3 in patients with cervical tumors of epithelial origin relapsing from first line treatment.
2. To determine disease free survival in patients treated with mAb Nimotuzumab hR3 for cervical tumors of epithelial origin when relapsing from first line treatment.
3. To determine the anti-tumoral response of mAb Nimotuzumab hR3 in patients with cervical tumors of epithelial origin relapsing from first line treatment.
4. To determine progression time of patients with cervical tumors of epithelial origin relapsing from first line treatment who were treated with mAb Nimotuzumab hR3 in combination with chemotherapy.
5. To evaluate the safety of mAb Nimotuzumab hR3 when treating patients with cervical tumors of epithelial origin relapsing from first line treatment in combination with Cisplatin/Vinorelbine chemotherapy.
6. To evaluate the appearing of HAMA response in patients treated with mAb Nimotuzumab hR3.
7. To evaluate the diminishing of associated symptoms in patients with cervical tumors of epithelial origin in relapse treated with mAb Nimotuzumab hR3.
8. To evaluate the quality of life of both groups using questionnaires QLQ C-30 and QLQ CX 24 for patients with cervical cancer (See appendixes).
9. To evaluate the toxicity using V3 Toxicity criteria.
10. To evaluate cardiac toxicity through MUGA or cardiac USG in both groups.
11. For feasibility purposes it will be conducted a MUGA and Rs MG only in Mexican patients to evaluate their cardiac function in order to compare both studies before and after clinical evaluation

Whenever possible, researcher shall perform a pre-treatment biopsy to assess the EGF-R expression and its characteristics using immunohistochemical techniques. EGFR expression will not constitute an inclusion criterion in this trial but will be correlated retrospectively with the antitumor clinical response of those patients on whom a pre-treatment biopsy was performed.

A QLQ-c30v3 test will be applied for it has the characteristic of evaluating the impact of the disease and its treatment on the patient's functioning in the physical, psychological and social areas. The QLQ Cx24 Questionnaire is a specific instrument for measuring the quality of life in patients with cervical cancer through different clinical phases.

TREATMENT

INDUCTION PHASE:

200 mg mAb Nimotuzumab will be administered once a week (12 weeks) in combination with a Platin based chemotherapy (Cisplatin/Vinorelbine) in cycles administered every 21 days (up to 6). Both therapies will be administered endovenously. Response will be assessed after the 3rd chemotherapy + mAb vs placebo cycle through physical examination, CAR, or MRI. IF THERE IS A PARTIAL RESPONSE OR STABLE DISEASE in line with RECIST, patient shall continue planned treatment until 6th CT + mAb vs placebo cycle is completed. In case of PROGRESSION, another treatment scheme should be considered according to researcher criteria. Following 6th Chemotherapy + mAb vs placebo cycle patient should be assessed again after 28 days through physical examination, MRI and CAT to measure lesions and through RECIST criteria. 6th cycle evaluation will be based on basal target lesions measured at the beginning of study. IF STABLE DISEASE OR ANTITUMORAL RESPONSE IS ESTABLISHED patient will continue to the next planned study phase. In the event of PROGRESSION, a second line chemotherapy should be considered. During second line chemotherapy evaluation, Nimotuzumab administration every 14 days will be maintained

FOLLOW-UP THERAPY:

In case of STABLE DISEASE or ANTITUMORAL RESPONSE (complete or partial), an mAb hR3 vs Placebo dose will be maintained every 14 days without chemotherapy after this concomitancy phase until patient shows progression. mAb Nimotuzumab hR3 will be administered endovenously in a 250 mL saline solution in 30 min. infusion ambulatory. Following drug administration, patient should remain in the health care institution for at least 4 hours in order to guarantee immediate adverse reactions detection and its appropriate treatment.

EVALUATION OF RESPONSE

Survival of patient will be determined from the moment of inclusion until death, for two years.

Therapeutic success will be considered to have occurred when the patient survives more than 10.5 months in the branch treated with mAb Nimotuzumab, or when the difference between both groups is not less than 4 months and that of the mAb group is not greater than 10.5 months.

Therapeutic failure will be considered to have occurred when the patient does not survive the 6.5 months that are habitually reported in the literature, which is the median survival of patients treated only with Platinum

IMAGE RESPONSE CRITERIA:

An evaluation of target lesions will be made (complete response, partial response, progressive disease, stable disease)

HAMA RESPONSE WITH ELISA

EGF-R EXPRESSION The EGF-R expression will be evaluated in the samples of tumors from the patients using Immunohistochemical techniques. The pre-inclusion EGFR expression will not constitute an inclusion criterion, but it will be correlated retrospectively with the antitumoral clinical response.

DETERMINATION OF KRAS, KI 65, P53. Evaluation of the QLQ- 30 and Cx24 questionnaires will be done in cycles 3 and 6 of the first line of chemotherapy, and in the 3rd and 6th cycles of the second line of chemotherapy.

ADVERSE EVENTS All adverse events during the trial will be documented in patient's file and in the report forms of each case. Every adverse event will be reported including the strat date, termination date, severity, and possible relation with the drug studied (occurrence of and AE, description of AE, intensisity of AE, casualty relation, attitude following AE)

Severity of adverse events will be evaluated according to the following taxonomy:

Serious adverse event (Grade 3): Event that threatens the life of patient. Hospitalization of patient is required with the possible interruption of the drug studied.

Moderate adverse event (Grade 2): Patient requires a symptomatic treatment to continue with her customary daily actvities. A more frequent evaluation is required until adverse event disappears.

Mild adverse event (Grade 1): Patient may continue with her daily activities and does not requiere complementary pharmacological treatment.

Characterization of Adverse Events Main researcher will evaluate each adverse event and will determine their relation with the drug being studied according to the following possible cases. He/she will record his/her evaluation in the Adverse Event Report.

0.- Unrelated The adverse event cannot be related to the use of the drug studied or there is no temporal or causal relation of the identified effect (other than the use of the drug studied)

1. - Possibly related There is a temporal association or the cause of the effect may be related with other ethiologies (probable causes). The relation with the drug studied cannot be excluded.
2. - Probably related There is a temporal association although there are other possible but not probable causes

Reporting of Adverse Events will be made as follows:

1. Report to the monitor no later than 24 hours when a patient is still being studied.
2. Reporting of adverse event within 30 days when the patient has finished the study.
3. A summary of the clinical history will be prepared including a detailed description of adverse events (regardless the adverse event might be associated or not to the drug or procedures of the study).
4. All serious adverse events shall be reported to the Institutional Ethic Committee and to the Research Host Hospital
5. A Report on Adverse Events will be made using the Health Secretariat format

A report will be delivered to the monitor to perform the pertaining actions.

Why Study Cardiac Function In different toxicities, cardiac toxicity was mentioned previously as one of the side effects of treatment with chemotherapy. In other studies, in which a molecular target directed against the VEG + chemotherapy has been studied, it has demonstrated cardiac toxicity, which makes it necessary to consider it.

Currently, the evaluation of cardiac function takes place through Nuclear Medicine and has been established as a safe, effective, and low-cost method. Basal, MUGA and ECG measurements will be made prior chemotherapy in cycle 6 of first line CT. In case of second line chemotherapies, measurements will be made in cycles 3 and 6.

The importance of quality of life means: good state of mental, physical, and social health in patients that survive the cancer (Brunner et al.1995). Patients treated with radiotherapy vs. surgery or both, in local advanced cervical cancer, demonstrate that they do not achieve the same quality of life two years after the treatment compared to the control group (Klee et al. 2000, Cull et al. 1993). The EORTC developed and validated a program in order to evaluate the quality of life of patients that suffer from cancer (above all, cervical and breast cancer) before and during the treatment. The QLQ-c30v 3 (Holzner et al. 2001, Fayer et al. 2002, Aaronson 1993), has the characteristic of evaluating the impact of the disease and its treatment on the patient's functioning in the following areas: physical, psychological, and social.

Recently, the QLQ Cx 24 questionnaire (Greimel et al. 2006) is a specific instrument for measuring the quality of life in patients with cervical cancer, validated by the EORTC. It has the capacity to assess quality of life in different clinical stages; it evaluates aspects of the female reproductive system, sex life, and the discomforts caused by the local treatment; it has a Cronbach Alfa coefficient of 72%-82%; the disadvantage is that this questionnaire must be self-evaluative, and the majority of our patients have to be helped due to the fact that 80% of our population has an incomplete primary school education.

Basal measurements will be made prior chemotherapy in cycle 3, then in cycle 6 of first line chemotherapy. In the case of second line chemotherapies, measurements will be made at the beginning of second line chemotherapy and in cycles 3 and 6 of such chemotherapy.

During follow-up, Questionnaires QLQ 30 and CX 24 will be preformed every 6 months during the first two years and afterwards, annually until completion of 5 years.

FOLLOW-UP Post-study follow-up visits will be made every 3 months during the first 2 years; every 4 months during third year; every 6 months in the following year, and later on, annually or until progression.

The information collected during that period will be as follows:

Limited clinical history and physical examination; performance status assessment including weight and tumor lesion measurements for lesions than can be measured through a physical examination or image studies: BH, QS, PFH; relapsing, progression or recurrence date.

Cardiac function will be assessed with MUGA every 6 months during the first year and later on, annually.

Evaluation of Questionnaires QLQ- 30 and Cx24 will be performed every 6 months during the follow-up and for the first twol years, and then, annually up to 5 years.

Blinding procedure and methods for code treatment opening and access. Main clinical researcher is the ultimate person responsible for the appropriate patient attention and he/she will determine if patient shall continue or not the treatment being researched in the event an adverse event appears bearing a risk to the life of patient.

In each clinical site, the researcher or pharmaceutical person responsible for the institution will be provided with sealed envelopes stating the treatment each patient is receiving. If a patient needs clinical management due to the presence of severe or unexpected adverse events related to the product being studied and for which it is required to know the treatment patient is receiving, randomization envelopes will be opened.

Opening the randomization envelope will only be justified when a severe or unexpected averse event is present. In that case, the procedure followed and explanations for that procedure shall be recorded on patient's clinical history.

Sealed envelopes containing the treatment assigned for each patient will be prepared by the designated person at the CIM Regulatory Affairs Department and he/she will also label the vials based on the randomized list stating the treatment each patient is receiving.

ELIGIBILITY:
Inclusion Criteria:

* Patients who grant their written consent to participate in the trial;
* With persistent or recurrent local and/or systemic cervical cancer with a measurable disease through physical examination, CAT, or MRI;
* Diagnosed 90 days after concluding administration of chemotherapy + radotherapy to pelvis or pelvic extended fields chemo-radiotherapy;
* Pathological report with epidermal carcinoma, adenocarcinoma, adenosquamous carcinoma and glassy cell carcinoma;
* ECOG Performance Status ≤2;
* Life expectancy >6 months;
* LVEF >50 (MUGA or ecocardiogram)
* Normal function of organs and of bone marrow defined by laboratory parameters.

Exclusion Criteria:

* Pregnant or breastfeeding patients;
* Small cells and/or neuroendocrine cervical cancer;
* Receiving other oncospecific drug under research;
* Allergy history to compounds of chemical or biological similar composition to the monoclonal antibody being evaluated or to chemotherapeutic agents;
* Intercurrent non controlled diseases including active infections, symptomatic congestive cardiac failure, unstable angina pectoris, cardiac arrhythmia, decompensated diabetes and psychiatric disorders.
* With a second tumor; except for those who have received appropriate treatment for skin carcinomas (basal or squamous).
* Previous or concomitant malignancy except for non-melanoma skin carcinoma.
* Social, family or geographic conditions that suggest a poor study compliance.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2010-07; Primary Completion 2014-05 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Overall survival | 11 months
  Patient's survival since inclusion until death.

SECONDARY OUTCOMES:
Illness free survival | 6 months
  Patient´s survival will be evaluated from the moment of complete response until progression.
Antitumoral Response | 6 months
  Treatement response or progression will be evaluated according to the new International Criteria from Response Evaluation Committee in Solid Tumors (RECIST) (EJC 2009; 45: 228-247). Antitumoral response will be evaluated from patient´s inclusion after second and sixth quemoterapeutic line, and latter, every 3 months until second year of follow up for each patient.
Progression free survival | 3 months
  Time after treatment in wich illness remains unprogressive. It will be evaluated through antitumoral response on cycles 3 and 6 of first line chemotherapy, and on line 2 and every 3 months through first 2 years of follow up.
Safety | Every 2 weeks for a period of 3 years
  Safety will be evaluated according to occurrence of any adverse event (AE) on patients. AE will be described, including duration, treatment applied, intensity, causality relationship, attitude followed in the pace of the apparence of the AE and result of the treatment applied to counteract the AE.

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Cancerología, México, Tlalpan, Mexico